CLINICAL TRIAL: NCT02727075
Title: Performance Value of Research of Occult Gastrointestinal Bleeding by Immunoassay in the Diagnostic Process of Iron Deficiency Anemia in Patients Over 75 Years
Acronym: STRATAGANEMIE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P140307; AOR14082 (Other: Department of Clinical Research & Development - APHP)
Record Dates: First submitted 2016-03-08; First posted 2016-04-04 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2021-02

CONDITIONS: Occult Gastrointestinal Bleeding
Keywords: Occult Gastrointestinal Bleeding; Iron Deficiency Anemia; Aged 75 Years and Older
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal Occult Blood Test
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to characterize the diagnostic performance of immunological testing of occult gastrointestinal bleeding in stool in the population aged over 75 years with iron deficiency anemia.

As secondary objectives, the study aims to:

* determine a threshold of positivity optimizing the immunoassay performance for the study population, in accordance with the probabilities of error (false positives, false negatives) and weights (defined by expert consensus) allocated to these errors.
* Assess the benefit of a double measure of bleeding (two stools) by immunoassay compared to a single measure.

DETAILED DESCRIPTION:
Immunological testing will be performed systematically for each patient.

Research of blood in fecal sample will be based on 2 methods: one based on a qualitative immunochromatographic method (such as HemSign4 technique, Servibio, France; or all other techniques used at AP-HP) and another quantitative immunoturbidimetric method (OC-Sensor, Eiken, Japan). They will be performed systematically with two fresh fecal samples for each patient, before coloscopy examination.

Treating physicians will not be provided with the testing result. The diagnosis of reference will be established by experts based on the result of explorations (colonoscopy, coloscanner) and the patient's progression, blinded to the result of immunoassay.

The intrinsic characteristics of the immunoassay (sensitivity, specificity...) will be determined with reference to this reference diagnosis, using a positivity threshold defined using expert consensus on the weights to be allocated to potential errors.

2 modeling scenarios (without vs with immunological testing) using decision trees based on prevalence and diagnostic performance observed and stochastic simulations.

ELIGIBILITY:
Inclusion Criteria:

* Physical status score 3 or 4, aged 75 and older patient, (patients under guardianship may be included).
* Iron deficiency anemia (Hb≤120 g/l for a woman or Hb≤130 g/l for a man), and nonregenerative anemia with reticulocytes <120 000/mm3.
* Patient who has indication for colonoscopy and / or colonography examination, whatever the results of gastroscopy if performed.
* Have a health insurance.
* Informed consent signed.

Exclusion Criteria:

* Hematemesis or melena
* Life expectancy inferior to 12 months
* Patient has difficulty in follow-up of study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 200 people at least 75 years old.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of immunological test with OC-SENSOR supplies | At baseline
  The immunological test with OC-SENSOR supplies is a quantitative determination of hemoglobin, the method of detection of lower gastrointestinal hemorrhagic lesions of older population with iron deficiency anemia.
  Sensitivity of the immunological test will be calculated statistically.
Specificity of immunological test with OC-SENSOR supplies | At baseline
  The immunological test with OC-SENSOR supplies is a quantitative determination of hemoglobin, the method of detection of lower gastrointestinal hemorrhagic lesions of older population with iron deficiency anemia.
  Specificity of the immunological test will be calculated statistically.
Likelihood ratios of immunological test with OC-SENSOR supplies | At baseline
  The immunological test with OC-SENSOR supplies is a quantitative determination of hemoglobin, the method of detection of lower gastrointestinal hemorrhagic lesions of older population with iron deficiency anemia.
  Likelihood rations of the immunological test will be calculated statistically.

SECONDARY OUTCOMES:
Diagnostic Performance | At baseline
  Diagnostic Performance of predictive equation incorporating all individual data will be calculated statistically.
Comparing scenarios using decision trees | At baseline
  Compare using modeling (decision trees) the causal efficiency (number of origins of bleeding detected / number of coloscopy-colonoscopy performed) of two scenarios: without (base case) and with the immunoassay to research occult bleeding in feaces (with one or two fecal samples).
Performance of the test when used with an optimized positivity threshold | At baseline
  Sensitivity, specificity and likelihood ratios of the immunological testing will be calculated statistically, when an optimized positivity threshold for the population under study is used, as a function of weights (defined by experts consensus) allocated to errors (false negative and false positive cases).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Lamarque, MD, PhD, Study Director — Service Hépato-Gastroentérologie, Hôpital Ambroise Paré
Locations (1):
- Service Hépato-Gastroentérologie, Hôpital Ambroise Paré, Boulogne-Billancourt, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No